CLINICAL TRIAL: NCT02131545
Title: A Single Dose Pharmacokinetic Study of Topical and Rectal Quetiapine Compared to Oral Quetiapine in Healthy Adults
Brief Title: Pharmacokinetic Study Comparing Topical, Rectal, and Oral Quetiapine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Jonathan G. Leung, Pharm.D., R.Ph., Psychiatric Clinical Pharmacist, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 14-000896
Record Dates: First submitted 2014-05-01; First posted 2014-05-06 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Dementia; Delirium
Keywords: quetiapine; pharmacokinetics; dementia; delirium; palliative care
MeSH Terms: conditions — Dementia; Delirium | interventions — Quetiapine Fumarate; Suppositories

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Quetiapine (Experimental): Quetiapine 25 mg
  Interventions: Drug: Quetiapine 25 mg gel applied topically; Drug: Quetiapine 25 mg tablet by mouth; Drug: Quetiapine 25 mg rectal suppository

INTERVENTIONS:
Drug: Quetiapine 25 mg gel applied topically — Quetiapine 25 mg gel applied topically; 9 serum quetiapine levels drawn over the course of 8 hours
  Other Names: Seroquel
Drug: Quetiapine 25 mg tablet by mouth — Quetiapine 25 mg tablet administered by mouth; 9 serum quetiapine levels drawn over the course of 8 hours
  Other Names: Seroquel
Drug: Quetiapine 25 mg rectal suppository — Quetiapine 25 mg suppository administered rectally; 9 serum quetiapine levels drawn over the course of 8 hours
  Other Names: Quetiapine
Drug: Quetiapine 25 mg gel applied topically — Quetiapine 75 mg gel applied topically every 4 hours for 24 hours; 6 serum quetiapine levels drawn over the course of 24 hours
  Other Names: Seroquel

SUMMARY:
Quetiapine, a second generation antipsychotic, is only available as oral tablets. However, topical and rectal formulations have been produced in compounding pharmacies. There is no data available suggesting that topical or rectal formulations provide serum levels similar to oral medication. In the clinical setting, when oral administration of quetiapine is not possible (for example, when a patient is extremely ill physically or mentally or both), clinicians and pharmacists have collaborated in such cases and have at times had to administer quetiapine compounded in other dosage formulations such as rectal or topical formulations. Despite clinical effectiveness of these other formulations, there are no available studies that have investigated blood levels of the drug other than the oral form. The investigators are therefore designing this pharmacokinetic study to evaluate the the systemic absorption of quetiapine in oral, rectal and topical formulations. If the investigators are able to demonstrate detectable levels from rectal and topical quetiapine formulations compared to the oral form, this knowledge will enhance clinical psychiatric practice by providing a more broad route of administration for quetiapine which is a commonly used drug for psychiatric symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult volunteers (18-65 years old) willing to undergo a general health screen consisting of blood pressure, heart rate, respiratory rate, height, weight, temperature, and electrocardiogram will be identified.
* The below parameters must be met to be consider an adult healthy to volunteer for inclusion in this study:
* Blood pressure less than 160/99 mmHg and greater than 105/50 mmHg

  * Heart rate between 50-100 beats per minutes
  * Respiratory rate between 10-30 breaths per minute
  * Temperature between 34 °C and 37.5°F
  * Corrected QT interval of < 470 msec
  * Liver function tests less than 1.5 times the upper limit of normal
  * Estimated creatinine clearance (estimated by Cockcroft Gault formulation) greater than 60 mL/min
  * Female participants will complete a urine pregnancy test that must result in a negative finding

Exclusion:

1. Allergy to quetiapine, Lipoderm or polyethylene glycol
2. Currently taking quetiapine
3. Pregnant, planning to become pregnant or breast feeding
4. Over or under 30% of ideal body weight
5. History of or active cardiovascular disease (except hypertension meeting the inclusion criteria for blood pressure), severe kidney disease (i.e. needing dialysis), or liver disease
6. History of schizophrenia, bipolar disorder, substance use disorders (but excluding nicotine use disorders and stable unipolar depression (See below))
7. Unstable unipolar depression, defined as hospitalization for depression within 1 year or changes to an antidepressant regimen within 6 months
8. History of seizure or seizure disorder
9. Parkinson's disease, Huntington's disease, tardive dyskinesia or other diagnosed movement disorder
10. History of/or active hematologic/oncologic illness
11. Dementia
12. Human Immunodeficiency Virus/Acquired Immunodeficiency Syndrome
13. History of organ transplant
14. History of gastric bypass
15. Contraindications for suppository administration
16. With Ostomy, chronic diarrhea
17. Diabetes, type 1 or type 2
18. Prolong corrected QT interval (>470 msec) or history of congenital long QT syndrome
19. Open wound(s) or unhealed wound(s) at topical medication application site (anterior forearm)
20. Active or latent tuberculous and currently prescribed pharmacotherapy treatments
21. Currently prescribed or taken with in the last 7 days, medications which have a known interaction with quetiapine or compound the risk of adverse events associated with quetiapine:

    * QTc prolonging medications:

      * Antipsychotics
      * Vaughan Williams Class IA, IB, IC, III antiarrhythmics
      * Anti-infective agents (excluding topical agents, oral penicillins, oral cephalosporins)
      * Antiemetics
      * Methadone
      * Cisapride
      * Cimetidine
      * Divalproex sodium/valproic acid
      * Tetrabenazine
      * Solifenacin
      * Tricyclic antidepressants
      * Tizanidine
      * Fingolimod
    * Increase quetiapine concentrations, not previously mentioned

      * Paroxetine
      * Fluoxetine
      * Fluvoxamine
      * Non-dihydropyridine calcium channel blockers (verapamil, diltiazem)
      * Tamoxifen
      * Cyclosporin (excluding ophthalmic formulation)
      * Nefazodone
    * Decrease quetiapine levels, not previously mentioned

      * Bosentan
      * Carbamazepine
      * Glucocorticoids
      * Modafinil
      * Primidone
      * St. John's wort
      * Barbiturates
      * Phenytoin
22. Vulnerable populations will be excluded (i.e. prisoners, wards of the state, emancipated minors, children, pregnant women)
23. Inability to receive telephone calls for the purpose of post-intervention follow-up
24. Inability or unwillingness of individual to give written informed consent
25. Non-English speaking populations

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Serum quetiapine levels after topical application (Visit 1) | 8 hours
  Areas under the curve versus time
Serum quetiapine levels after oral administration (Visit 2) | 8 hours (no sooner than 72 hours from end of visit 1)
  Areas under the curve versus time
Serum quetiapine levels after rectal administration (Visit 3) | 8 hours (no sooner than 72 hours from end of visit 2)
  Areas under the curve versus time

SECONDARY OUTCOMES:
Serum quetiapine levels after topical administration over 24 hours | 24 hours
  Topical quetiapine applied every 4 hours for 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Leung, PharmD, RPh, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided